CLINICAL TRIAL: NCT05520346
Title: Testing a Device for Automatically TRacking Urine and STool in an Inpatient HCT Setting (Project TRUST)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00107848
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Fluid Output
Keywords: toilet device
MeSH Terms: interventions — Bathroom Equipment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Device (Experimental): Patients use toilet device to measure fluid output and self-report event types
  Interventions: Device: Electronic Device for Toilet
- Control (No Intervention): Collection in standard hats + nurses visually assessing fluid volumes

INTERVENTIONS:
Device: Electronic Device for Toilet — Device will be installed on toilet of patients will in hospital to measure all waste output.
  Arms: Device

SUMMARY:
The purpose of this study is to determine whether a prototype toilet device that we have developed can accurately and automatically track human fluid output from renal and gastrointestinal systems in the hospital. The device includes components that can be outfitted onto existing toilets.

In this study, participants hospital room will be outfitted with the prototype toilet device. Participants will use the toilet as usual throughout the duration of their inpatient stay. Sometimes output will be measured by the device, and other times output will be measured manually by nurses.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo an allogeneic or autologous hematopoietic stem cell transplant for any cancer or non-cancer illness through the Duke ABMT clinic
* Age 18-80 years
* Karnofsky Performance Scale KPS ≥ 70
* Able to read/write English

Exclusion Criteria:

* Inability to use toilet device due to physical constraints, e.g. waste excreted through stoma or catheter
* Physician recommendation that patient does not use standard urine/stool collection hat during days 1-2 of HCT conditioning

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean absolute error of urine volume (in mL) as measured by device compared to standard of care nurse assessment | Up to 14 days

SECONDARY OUTCOMES:
Correlation between daily patient fluid balance (difference between fluid input and output in mL) as measured by device measurements or standard of care nurse assessment and the change in daily weight | Up to 14 days
Mean absolute error of urine volume (in mL) as measured by device | Up to 14 days
Time (in mins) spent handling/recording patient waste | First 3 days of patient's HCT conditioning
Levels of chemotherapy drugs detectable on room surfaces as measured by surface testing | First 3 days of patient's HCT conditioning
Time (in mins) between nurse logging of patient urination in electronic medical records and device-based logging of patient urination | Up to 14 days
Percent device can correctly identify diarrhea events | Up to 14 days
Percent of patients who indicated device satisfaction as measured by patient survey | Day 3 of HCT conditioning
Percent of nurses who perceived lower chemotherapy exposure as measured by survey | After transition to Stage 2 - about 3 days after patient begins HCT conditioning
Percent of nurses who indicated device satisfaction as measured by nurse survey | After transition to Stage 2 - about 3 days after patient begins HCT conditioning
Number of patient falls as measured by patient report | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Chenyu Lin, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No